CLINICAL TRIAL: NCT07272824
Title: Usability Study of Gestational and 6 Months Postpartum Weight Management Program - Hope D
Brief Title: Usability Study of Gestational and Postpartum Weight Management Program
Acronym: Hope-D_Use
Status: Recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Collaborators: Hospital District of Helsinki and Uusimaa (Other); University of Turku (Other); University of Helsinki (Other)
Responsible Party: Sponsor
Other Study IDs: Hope-D usability study
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy; Postpartum; Obese Pregnant Women; Weight Management; Digital Intervention; Usability
Keywords: Hope-D; digital pathway; Gestational weight management; Postpartum weight management; gestational weight management plan; coaching

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Usability of digital pathway, general/individual weight management plan and group/individual coachin: The participants will evaluate the digital pathway with a general and an individual gestational and 6 months postpartum weight management plan and group as well as individual coaching provided by a trained study nurse.

SUMMARY:
The principal aim of this study is to evaluate the usability of the Hope-D gestational and 6 months postpartum weight management program. We will evaluate the usability, functionality, and acceptability of the developed Hope-D weight management program that includes digital pathway for weight management, general or individual weight management plan and individual or group coaching for weight management from pregnancy to 6 months postpartum.

DETAILED DESCRIPTION:
The usability of the digital pathway will be evaluated through a one-week user test among up to 30 pregnant women, who have prepregnancy BMI at least 30 kg/m2.

Participants will use the Health Village digital pathway for gestational and 6 months postpartum weight management, after which they will take part in semi-structured interviews conducted via Microsoft Teams and complete the System Usability Scale (SUS) questionnaire assessing perceived acceptability and usability.

All interviews will be audio-recorded, transcribed verbatim, and analyzed qualitatively.

Participants will report whether they accessed the pathway via mobile phone or computer and evaluate the technical usability, including ease of login, fluency of navigation, functionality of links, and the overall visual design.

The content of the digital pathway will be assessed in terms of relevance, usefulness, completeness, and clarity. Participants will be asked whether all key topics were covered, which elements were most beneficial or motivating, and whether the content was appropriate for both the gestational and postpartum periods.

All participants will provide feedback on the weight management plan. Participants will review the general plan and the individual plan. Feedback will address the perceived suitability of the plan to support gestational and postpartum weight management, appropriateness of the six-month postpartum evaluation point, and the feasibility of presenting the plan in the digital maternity card.

All participants will evaluate the group coaching component. After reviewing the session themes, they will assess the added value of group coaching, appropriateness of session content and timing, complementarity to standard care, and preferences for individual coaching.

Similarly, participants will evaluate the individual coaching component, assessing its added value, appropriateness of content and timing, complementarity to standard care, and potential preference for group-based coaching.

ELIGIBILITY:
Inclusion Criteria:

* General pregnant women with prepregnancy BMI at least 30 kg/m2
* Competence in using the digital care pathway and electronic maternity card

Exclusion Criteria:

- Significant difficulty in cooperating (e.g. inadequate Finnish language skills)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gestational and postpartum weight management can be studied only in pregnant women.
Study Population: Pregnant women in the wellbeing services county of Southwest Finland, Turku area
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
The basic version of Hope-D program has been developed | 1 week
  The aim of the Hope-D program is to develop a standardized model for gestational and postpartum weight management. The basic version of the Hope-D program will be considered ready for implementation in the subsequent intervention study once all sections of the System Usability Scale (SUS) reach a score above 68 within the same development period (sprint).
  The SUS is a widely used, reliable, and valid instrument for evaluating the usability of various technologies, including digital products, systems, and services. It comprises ten statements rated on a five-point Likert scale, where 1 indicates strong disagreement and 5 indicates strong agreement. The total SUS score ranges from 0 to 100, with higher scores indicating better perceived usability. The SUS questionnaire has been translated into Finnish and is available for use free of charge.

SECONDARY OUTCOMES:
Usability of gestational and postpartum digital pathway for weight management | 1 week
  General technical questions will address the usability aspects and general thematic questions, e.g., motivation to manage weight during and after pregnancy with a digital pathway for weight management. Participants' responses will provide qualitative insights to guide the further development of the Hope-D program. The responses will not be quantitatively scored, as there are no right or wrong answers. Instead, the data will be analyzed using qualitative content analysis. Themes and issues that emerge most frequently across interviews will be considered the most relevant usability concerns and will be given higher priority in the development guidelines than those mentioned only occasionally.
Usability of gestational and postpartum general and individual weight management plan | one week
  The general interview questions focus on the visibility and relevance of the weight management plan, the types of support perceived as motivational, clarity of goal-setting, and the appropriate timing for initiating and continuing weight management during pregnancy and in the postpartum period.
  Participants' responses will inform the development of the Hope-D application. The data will be analyzed qualitatively; responses will not be scaled or scored, and there are no right or wrong answers. Recurring themes identified across multiple interviews will be considered indicative of common needs and prioritized accordingly in the development of the application guidelines. Themes mentioned in single interviews will also be noted but will receive lower priority in the guideline development process.
Usability of group and individual coaching sessions | one week
  The general interview questions explore whether group or individual coaching sessions add value to the digital pathway for weight management and general weight management plan. Themes include the perceived usefulness of coaching, optimal number and spacing of sessions, and the suitability of specific topics for either individual or group coaching formats. The answers of participants give investigators the guidelines for the development of Hope-D application. The answers themselves won't be scored; there aren't wrong or correct answers. Answers which repeat most commonly in the interviews are the most common issues and they will have higher priority in the guideline than answers which arise only in one interview.

CONTACTS AND LOCATIONS:
Overall Officials: Kaarin Mäkikallio, Study Director — The wellbeing services county of Southwest Finland
Locations (1):
- The wellbeing services county of Southwest Finland, Turku, Finland, Finland

IPD SHARING:
Plan to Share IPD: No
EU GDPR restricts data sharing